CLINICAL TRIAL: NCT02313779
Title: Nonconscious Affective and Physiological Mediators of Behavioral Decision Making Study 3
Brief Title: Meditation and Decision Making Study III
Acronym: MDMS3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara L. Fredrickson, PhD (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Barbara L. Fredrickson, PhD, Nonconscious Affective and Physiological Mediators of Behavioral Decision Making Study 3, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 12-2428; R01AT007884-01 (NIH)
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Meditation
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Neutral (Placebo Comparator): Reading passage about brain function which is masked as a news article.
  Interventions: Behavioral: Lovingkindness Meditation (LKM); Behavioral: Mindfulness Meditation
- Lovingkindness Meditation (LKM) (Experimental): Lovingkindness guided meditation experienced in the laboratory and 6 additional LKM meditations taken home on the iPod.
  Interventions: Behavioral: Lovingkindness Meditation (LKM)
- Mindfulness Meditation (Placebo Comparator): Mindfulness guided meditation experienced in the laboratory and 6 additional Mindfulness meditations taken home on the iPod.
  Interventions: Behavioral: Mindfulness Meditation
- Positivity (Experimental): Reading passage about prioritizing positive emotions which is masked as a news article.
  Interventions: Behavioral: Lovingkindness Meditation (LKM); Behavioral: Mindfulness Meditation

INTERVENTIONS:
Behavioral: Lovingkindness Meditation (LKM) — Compassionate behavior training (REVISE)
  Arms: Lovingkindness Meditation (LKM); Neutral; Positivity
Behavioral: Mindfulness Meditation
  Arms: Mindfulness Meditation; Neutral; Positivity

SUMMARY:
The overarching goal of the proposed research is to investigate the role of emotions in facilitating successful lifestyle change, defined as healthy behavioral decisions repeated daily, or near daily.

Participants are asked to make two lab visits during the course of four weeks to complete electronic questionnaires, be monitored for psychophysiological activity (e.g. heart rate, blood pressure, respiration), and listen to a guided meditation audio track. Additionally, between the two visits participants will be asked to complete weekly surveys that ask about daily meditation practice (outside of the lab) and general emotions.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in written and spoken English, with a high school reading level
* Willingness or interest in learning to meditate
* Computer literate with internet access

Exclusion Criteria:

* Individuals who are able to read Chinese logographs
* Individuals who have or have had a regular meditation practice, defined as having attended a 6-week or longer meditation class, practicing meditation at least 3 days a week for up to 6-weeks.
* Individuals with allergies to adhesive materials

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in positive emotions (as measured by the Modified Daily Emotions Scale) | Baseline and Weeks 1, 2, and 3
  Modified Daily Emotions Scale (mDES) - This measure of explicit positive affect has been successfully used by the PI in multiple studies to detect changes in positive emotion. Previous work by the PI found that Cronbach's alpha coefficient for the mDES positive emotion composite variable was 0.93 in sample of mid-life community adults similar to those anticipated for this study.
Change in nonconscious incentive salience (as measured by the Affect Misattribution Procedure) | Baseline and Weeks 1, 2, and 3
  Affect Misattribution Procedure (AMP) - This measure of nonconscious incentive salience has acceptable internal consistency for an indirect measure of affect (.69 - .90) and has been found to predict judgments and behavioral outcomes above and beyond self-report measures.
Changes in meditation time | Weeks 1, 2, and 3
  Self-reported meditation time recorded daily and weekly. In addition, meditation track play times will be recorded from the iPod.

SECONDARY OUTCOMES:
Cardiac Vagal Tone | Baseline
  This measure of parasympathetic control over the heart has been positively associated with both emotional and social functioning. Previous work by the PI's team has found that baseline vagal tone predicts increased positive response to lovingkindness meditation (LKM), and that LKM in turn increases vagal tone.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Fredrickson, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC PEP Lab, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Fredrickson BL, Cohn MA, Coffey KA, Pek J, Finkel SM. Open hearts build lives: positive emotions, induced through loving-kindness meditation, build consequential personal resources. J Pers Soc Psychol. 2008 Nov;95(5):1045-1062. doi: 10.1037/a0013262. PMID 18954193
- [Background] Carmody J, Baer RA, L B Lykins E, Olendzki N. An empirical study of the mechanisms of mindfulness in a mindfulness-based stress reduction program. J Clin Psychol. 2009 Jun;65(6):613-26. doi: 10.1002/jclp.20579. PMID 19267330
- [Background] Johnson KJ, Waugh CE, Fredrickson BL. Smile to see the forest: Facially expressed positive emotions broaden cognition. Cogn Emot. 2010 Feb 19;24(2):299-321. doi: 10.1080/02699930903384667. PMID 23275681
- [Background] Payne BK, Cheng CM, Govorun O, Stewart BD. An inkblot for attitudes: affect misattribution as implicit measurement. J Pers Soc Psychol. 2005 Sep;89(3):277-93. doi: 10.1037/0022-3514.89.3.277. PMID 16248714